CLINICAL TRIAL: NCT05525455
Title: A Phase 1/2, First-in-human Study of the Safety, Pharmacokinetics, and Preliminary Anti-tumor Activity of TT-816 As Monotherapy or in Combination with a PD-1 Inhibitor in Patients with Advanced Cancers (SEABEAM) (MK3475-E88)
Brief Title: TT-816 As Monotherapy or in Combination with a PD-1 Inhibitor in Patients with Advanced Cancers (SEABEAM) (MK3475-E88)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company operational decision. Decision to stop study is not due to safety or efficacy concerns.
Sponsor: Teon Therapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SEABEAM
Record Dates: First submitted 2022-08-22; First posted 2022-09-01 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2023-10

CONDITIONS: Advanced Cancer; Advanced Solid Tumor; Cancer; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose and dose-expansion of TT-816 administered as a single agent or in combination with a PD-1 inhibitor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single agent TT-816 (Experimental): Escalating doses followed by expansion targeting advanced cancers
  Interventions: Drug: TT-816
- Combination TT-816 plus a PD-1 inhibitor (Experimental): Escalating doses followed by expansion targeting advanced cancers
  Interventions: Drug: TT-816; Drug: A PD-1 inhibitor

INTERVENTIONS:
Drug: TT-816 — TT-816 is a novel, oral cannabinoid CB2 receptor antagonist acting as an immune checkpoint inhibitor for the treatment of a broad range of solid tumors
Drug: A PD-1 inhibitor — Programmed death receptor-1 (PD 1)-blocking antibody
  Arms: Combination TT-816 plus a PD-1 inhibitor

SUMMARY:
A first-in-human study using TT-816 as a single agent and in combination with a PD-1 inhibitor in advanced cancers.

DETAILED DESCRIPTION:
This is an open-label, Phase 1/2, first-in-human (FIH), multiple ascending dose and dose-expansion study of TT-816 administered as monotherapy and in combination with a PD-1 inhibitor. Phase 1 will define the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of TT-816 and of combination therapy that can be advanced to Phase 2. Phase 2 will define the preliminary efficacy of these regimens in the setting of advanced solid tumors with high unmet medical needs including Non-Small Cell Lung Cancer (NSCLC), Ovarian Cancer and Renal Cell Carcinoma (RCC).

ELIGIBILITY:
All patients, regardless of phase or cohort, must meet the following criteria to be eligible for participation in the study:

1. Age ≥ 18 years old on day of signing informed consent.
2. Phase 1 - Cohorts 1m and 1p:

   1. Patients histologically or cytologically documented, locally advanced or metastatic solid tumor.
   2. Has disease that is measurable by RECIST 1.1 or evaluable disease. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
   3. Disease progression confirmed by imaging or other objective evidence after having received standard treatment; or patients with refractory solid tumors who cannot tolerate standard treatment or have contraindications to standard treatment.
3. Phase 2 - Non-Small Cell Lung Cancer (NSCLC) (Cohorts 2m1 and 2p1):

   1. Patients with histologically or cytologically documented Stage IV NSCLC not amenable to curative surgery or radiation.
   2. Patients enrolling in cohort 2m1 must have progressed on a platinum containing chemotherapy or an anti PD-1 pathway therapy. Patients enrolling in cohort 2p1 must have progressed on or after a platinum containing chemotherapy and an anti-PD-1 pathway therapy.
   3. Patients must not have known gene alterations (such as EGFR, ALK, ROS-1, or RET) at the time of screening.
4. Phase 2 - Ovarian Cancer (Cohorts 2m2 and 2p2):

   1. Patients with histologically or cytologically confirmed ovarian epithelial cancer.
   2. Evidence of progressive disease (PD) on or within 6 months of a platinum (cisplatin or carboplatin) regimen.
   3. At least 1 prior regimen must have contained a platinum-taxane combination.
5. Phase 2 - Renal Cell Carcinoma (Cohorts 2m3 and 2p3):

   a. Histologically confirmed locally advanced or metastatic clear cell renal cell carcinoma that has progressed during or after at least two prior therapeutic regimens which must include vascular endothelial growth factor (VEGF)-targeted therapy and checkpoint inhibitor therapy or that has otherwise failed such therapies and is measurable disease per RECIST 1.1 criteria.
6. Phase 2 - Cohorts 2m and 2p: Have disease that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
8. Expected life expectancy of greater than 12 weeks per the Investigator.
9. Capable of swallowing a medication in full tablet form, without the need to crush the medication.
10. Adequate coagulation function defined as the following at screening:

    1. Prothrombin time (PT) and International Normalized Ratio (INR) < 1.5 times the ULN
    2. Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 times the ULN unless undergoing anticoagulation therapy with warfarin
11. Female patients must have a negative urine pregnancy test at screening (within 72 hours of first dose of study drug) if of childbearing potential or be of non-childbearing potential. If the urine test is positive or cannot be confirmed as negative, then the patient must have a serum pregnancy test (β-human chorionic gonadotropin [β-HCG]). Non-childbearing potential is defined as (by other than medical reasons): a. ≥ 45 years of age and has not had menses for greater than 1 year b. Amenorrheic for ≥ 2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone (FSH) value in the postmenopausal range at screening, c. Status post hysterectomy, oophorectomy, or tubal ligation
12. Female patients of childbearing potential (FOCP) must agree to abstain from heterosexual intercourse or use a highly effective form of contraception from the time of informed consent, during the study, and for 4 months following the last dose of study drug(s).
13. Male patients with partners of childbearing potential must agree to abstain from sexual intercourse or to use a highly effective form of contraception from the time of informed consent, during the study, and for 4 months following the last dose of study drug(s).
14. The patient (or legally authorized representative, if applicable) provides written informed consent for the study.
15. Willing and able to provide blood samples prior to the start of this study.

    For Phases 1m and 2m, patients must meet the following criteria to be eligible for participation in the study:
16. Adequate bone marrow function defined as:

    a. Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3 b. Platelet count ≥ 75,000 cells/mm3 c. Hemoglobin ≥ 8.0 g/dL
17. Adequate renal and hepatic function defined as:

    1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 4 times the upper limit of normal (ULN)
    2. Total bilirubin ≤ 1.5 times the ULN. If total bilirubin is > 1.5 times the ULN, then direct bilirubin must be less than or equal to the ULN. For patients with liver metastases or Gilberts Syndrome total bilirubin ≤ 2.5 times the ULN
    3. Creatinine clearance (CrCl) ≥ 60 mL/min calculated per institutional standard

    For Phases 1p and 2p, patients must meet the following criteria to be eligible for participation in the study:
18. Adequate bone marrow function defined as the following at screening and confirmed within 10 days prior to the start of study drug:

    a. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3 b. Platelet count ≥ 100,000 cells/mm3 c. Hemoglobin ≥ 9.0 g/dL (this criterion must be met without packed red blood cell (pRBC) transfusion within the prior 2 weeks. Patients can be on stable dose of erythropoietin (≥ approximately 3 months)).
19. Adequate renal and hepatic function defined as the following at screening and confirmed within 10 days prior to the start of study drug:

    1. AST and ALT ≤ 2.5 times the ULN (≤ 5 times the ULN for patients with liver metastases)
    2. Total bilirubin ≤ 1.5 times the ULN. If total bilirubin is > 1.5 times the ULN, then direct bilirubin must be less than or equal to the ULN. For patients with liver metastases or Gilberts Syndrome total bilirubin ≤ 2.5 times the ULN.
    3. Creatinine clearance (CrCl) ≥ 60 mL/min calculated per institutional standard. Glomerular filtration rate (GFR) may be used in place of creatinine or CrCl and must be > 1.5 times the institutional ULN.
20. For those patients with prior disease progression on treatment with an anti-PD1/L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies, the PD-1 treatment progression must meet all of the following criteria: a. Has received at least 2 doses of an approved anti-PD-1/L1 mAb. b. Has demonstrated disease progression (PD) after PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than four weeks from the date of the first documented PD, in the absence of rapid clinical progression.

    c. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

    i. Progressive disease is determined according to iRECIST. ii. This determination is made by the investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.

Exclusion Criteria:

All patients, regardless of phase or cohort, who meet any of the following criteria will not be eligible for participation in the study:

1. Received another systemic anticancer therapy including investigational agents within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose of study drug. Note: Patients must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Patients with ≤ Grade 2 neuropathy may be eligible. Patients with endocrine-related AEs ≤ Grade 2 requiring treatment or hormone replacement may be eligible.
2. Received radiotherapy within 2 weeks prior to the first dose of study drug or palliative radiation therapy within 1 week prior to the first dose of study drug.
3. Have another primary malignancy that is progressing, has required active treatment within the last 3 years, or has not been treated with curative intent within the last 3 years (discuss with Medical Monitor). Patients with carcinoma-in-situ that has been treated successfully more than 3 years prior to screening, non-metastatic cutaneous basal cell or squamous cell carcinoma, or non-muscle invasive bladder cancer are not excluded.
4. Have untreated central nervous system (CNS), epidural tumor or metastasis, or brain metastasis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (repeat MRI or CT with contrast should be performed during study screening), clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
5. Major surgical procedures within 4 weeks (28 days) of the first dose of study drug. If the patient had major surgery, the patient must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study drug.
6. Patients previously enrolled on this study and received at least one dose of study drug.
7. Is currently participating in or has participated in a study of an investigational agent or therapy, or has used an implantable investigational device within 4 weeks prior to the first dose of study treatment. Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
8. Have a QT interval corrected (QTc) prolongation to > 470 milliseconds (ms) at screening based on a 12-lead electrocardiogram (ECG) in triplicate using the Fridericia formula (QTcF): QTc = QT / RR 1/3.
9. Patients on concomitant medications that increase or possibly increase the risk of QTc prolongation and/or induce Torsades de Pointes, including antifungals, antibiotics, antipsychotics, antiemetics, antiarrhythmics, and antineoplastic medications.
10. Patients on proton pump inhibitors (PPIs) who cannot switch to H2 inhibitors (or cannot stop PPI therapy entirely) at least 3 days before their first dose of TT-816 study drug for the duration of the study. See protocol Section 5.2 for permissible usage of H2 inhibitors during the study.
11. Have received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Administration of killed vaccines are allowed.
12. Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
13. Have a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease
14. Have significant, uncontrolled, or active cardiovascular disease, including, but not restricted to:

    1. Myocardial infarction (MI) or unstable angina within 6 months before the first dose of study drug.
    2. History of an arterial thrombotic event, stroke, or transient ischemia attack within 12 months prior to first dose of study drug
    3. Symptomatic congestive heart failure (New York Heart Association classes II-IV) within 6 months before the first dose of study drug
    4. A cardiac arrhythmia that requires treatment within 6 months before the first dose of study drug
15. Patients with evidence of an active infection requiring intravenous (IV) antibiotics within 7 days prior to the first dose of study drug.
16. Patients with active uncontrolled bleeding, or a bleeding diathesis within 7 days prior to the first dose of study drug.
17. Patients with serious or non-healing wound, fistula, skin ulcer, or non-healing bone fracture within 7 days prior to the first dose of study drug.
18. Patients with known history of human immunodeficiency virus (HIV) infection. Note: No HIV testing is required unless patient history of HIV is unknown or if mandated by local health authority.
19. Patients with a known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus infection (defined as HCV RNA [qualitative] is detected). Note: No testing for Hepatitis B and Hepatitis C is required unless patient history of Hepatitis B or Hepatitis C is unknown or if mandated by local health authority.
20. Pregnant or breastfeeding or plans to become pregnant during the study.
21. Patients unwilling or unable to follow protocol requirements, including any known psychiatric or substance use disorder that would interfere with the patient's ability to comply with the requirements of the study.
22. Have a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient to participate, in the opinion of the Investigator.

    There are no additional exclusionary criteria specific to participation in Phases 1m and 2m.

    For Phases 1p and 2p, patients who meet any of the following criteria will not be eligible for participation in the study:
23. Have severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
24. Have any history of radiation pneumonitis. Note: Patients must have recovered from all radiation-related toxicities and not require corticosteroids.
25. Have received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), and was discontinued from that treatment due to an irAE.
26. Have had an allogeneic tissue/solid organ transplant.
27. For patients with NSCLC, have received radiation therapy to the lung that is >30Gy within 6 months of the first dose of trial treatment.
28. Have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) - (Phase 1) | 3 years
  Incidence of adverse events (AEs) and serious adverse events (SAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Incidence and nature of dose-limiting toxicities (DLTs) - (Phase 1) | up to 21 days
  Incidence and nature of DLTs within a 3+3 trial design
Changes from baseline in clinical safety laboratory values and vital signs | 2 years
  Changes from baseline in clinical safety laboratory values and vital signs
MTD or RP2D of oral TT816 - (Phase 1m) | 1 year
  The Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) of oral TT-816 as monotherapy (Phase 1m)
MTD or RP2D of oral TT816 - (Phase 1p) | 1 year
  The Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) of oral TT-816 in combination with a PD-1 inhibitor (Phase 1p)
Efficacy assessments according to RECIST 1.1 (Phase 2) | 3 years
  Overall Response Rate. Scale: confirmed Complete response (CR) or Partial response (PR), Duration of Response (DOR), and Disease Control Rate (DCR).

SECONDARY OUTCOMES:
Objective response rate (ORR). - (Phase 1) | 3 years
  Efficacy assessments according to RECIST 1.1. Objective Response Rate (ORR) Scale: Complete response (CR), Partial response (PR)
Disease control rate (DCR) (Phase 1) | 3 years
  Disease control rate (DCR)
Duration of response (DOR) (Phase 1) | 3 years
  Duration of Response (DOR)
Progression-free survival (PFS) (Phase 1) | 3 years
  Progression-free survival (PFS)
Overall survival (OS) (Phase 1) | 3 years
  Overall survival (OS).
PK (Cmax) of TT-816 - (Phase 1) | 2 years
  Noncompartmental Pharmacokinetic (PK) parameters of TT-816 including the maximum plasma concentration (Cmax )
PK (AUC) of TT-816 - (Phase 1) | 2 years
  Noncompartmental PK parameters of TT-816 including area under the plasma concentration-time curve (AUC)
Incidence of AESIs - (Phase 2) | 3 years
  Incidence of AEs of special interest
Incidence of AEs and SAEs - (Phase 2) | 3 years
  Incidence of AEs and SAEs graded according to the NCI CTCAE v5.0
PK (Cmax) of TT-816 - (Phase 2) | 2 years
  Noncompartmental PK parameters of TT-816 including the maximum plasma concentration (Cmax )
PK (AUC) of TT-816 - (Phase 2) | 2 years
  Noncompartmental PK parameters of TT-816 including area under the plasma concentration-time curve (AUC)
PFS and OS - (Phase 2) | 3 years
  Progression Free Survival (PFS) and Overall Survival (OS)

OTHER OUTCOMES:
Food effects on PK parameters (Phase 2) | 2 years
  Comparison of PK parameters of TT-816 when given with food compared to fasted conditions to see if food or fasted conditions change the concentration of TT-816 in the blood.
Molecular analysis of patient tissue (Phase 1 and Phase 2) | 2 years
  Molecular analysis of patients' tumor and plasma may include, but is not limited to IHC
Molecular analysis of patient tissue (Phase 1 and Phase 2) | 2 years
  Molecular analysis of patients' tumor and plasma may include, but is not limited to mRNA expression.
Molecular analysis of patient tissue (Phase 1 and Phase 2) | 2 years
  Molecular analysis of patients' tumor and plasma may include, but is not limited to ctDNA and mutations.
Molecular analysis of patient tissue (Phase 1 and Phase 2) | 2 years
  Molecular analysis of patients' tumor and plasma may include, but is not limited to CB2R gene expression
Molecular analysis of patient tissue (Phase 1 and Phase 2) | 2 years
  Molecular analysis of patients' tumor and plasma may include, but is not limited to Circulating immune cells in peripheral blood mononuclear cells (PBMCs)
Molecular analysis of patient tissue (Phase 1 and Phase 2) | 2 years
  Molecular analysis of patients' tumor and plasma may include, but is not limited to Plasma cytokines
Tumor assessments (Phase 1 and Phase 2) | 2 years
  Tumor assessments based on iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Teon Clinical Development, Study Director — Teon Therapeutics, Inc.
Locations (5):
- United States (5):
  - Teon Investigational Site, Nashville, Tennessee
  - Teon Investigational Site, Austin, Texas
  - Teon Investigational Site, San Antonio, Texas
  - Teon Investigational Site, West Valley City, Utah
  - Teon Investigational Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No